CLINICAL TRIAL: NCT07387341
Title: Long-acting Spatial Emanators / Repellents (LASER) vs Indoor Residual Spraying (IRS) in Western Kenya: a Cluster-randomised Trial
Brief Title: Long-acting Spatial Emanators / Repellents (LASER)
Acronym: LASER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Institute of Tropical Medicine, Belgium (Other); Radboud University Medical Center (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 101190818
Record Dates: First submitted 2025-12-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Malaria Transmission; Malaria Prevention; Malaria
Keywords: spatial repellents; spatial emanators; Indoor Residual Spraying; Kenya
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Two interventions will be evaluated in this trial: (i) LASER (intervention #1) and (ii) IRS with pirimiphos-methyl (intervention #2), as compared to standard of care (control) in a parallel 1:1:1 open label cluster randomised trial . All clusters will receive standard malaria control interventions, including LLINs distributed by the Kenyan NMCP and malaria vaccines (when and where these are deployed).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LASER (Experimental)
  Interventions: Device: Guardian
- IRS (Experimental)
  Interventions: Device: IRS with Pirimiphos - methyl
- Standard control (No Intervention)

INTERVENTIONS:
Device: Guardian — The SC Johnson long-acting product (Guardian™) is a vapor releasing product (VP) formed from a polyester (PET) mesh substrate carrier dosed with 2,500 mg of transfluthrin per unit (CAS No. 118721-89-3). Transfluthrin is a type I synthetic pyrethroid that acts through modulation of nerve axon sodium channels, causing neurotoxicity in insects. The product is intended to be used as spatial emanator for the control of mosquitoes. The insecticide emanates from the product and subsequently kills or disrupts the biting behaviour of the surrounding vector population. The LASER product will be procured locally from the SC Johnson factory in Nairobi, Kenya (SC Johnson).
  Arms: LASER
Device: IRS with Pirimiphos - methyl — In clusters that are randomised to the IRS arm, IRS will be carried out using pirimiphos-methyl (Actellic®300CS) manufactured by Syngenta, an organophosphate insecticide that is registered for use in Kenya and has demonstrated effectiveness in malaria vector control. The product will be obtained directly from Syngenta to ensure quality and authenticity, with proper documentation and chain of custody maintained throughout the procurement and storage process.
  Arms: IRS

SUMMARY:
Malaria is a major problem in western Kenya, particularly around Lake Victoria. Whilst current prevention methods like bed nets and vaccines help to reduce malaria burden, additional tools are needed to better protect communities from malaria. The investigators will test a new technology called LASER Guardian™, which are devices that release chemicals to keep mosquitoes away from homes. The investigators will conduct a large study involving 69 villages in western Kenya over two years. Each village will be randomly chosen to receive one of three approaches: the new LASER devices, indoor residual spraying with insecticide (a method already known to work), or the standard prevention methods currently used. All villages will continue to receive the usual malaria prevention tools provided by the Kenyan government, including bed nets and vaccines. In villages receiving LASER, the investigators will install 2-3 small device inside structures once a year for two years. In villages receiving IRS, the investigators will spray the inside walls of homes with insecticide once a year for two years. The investigators want to find out if the LASER devices can reduce malaria better than current methods alone, and whether they work as well as indoor spraying. To do this, the investigators will carry out surveys of the community every six months over two years (four rounds in total), testing about 4,485 children between ages 1 and 15 from approximately 3,450 households in each survey to see how many have malaria. The investigators will also work with local health clinics to track malaria cases, study mosquitoes to understand how the interventions affect them, talk with community members about their experiences, and calculate the costs of these different approaches. This study will help us understand whether LASER tool can effectively protecting against malaria in Kenya and other African countries where malaria is common.

ELIGIBILITY:
The inclusion criteria are:

1. Child aged 1-15 years
2. Usual resident (a person who has been residing in the survey area for at least the past 4 months) who was present in the sampled household on the night before the survey
3. Agreement of adult or parent/guardian (of children) to provide informed consent
4. Agreement of child aged 12 years or older to provide assent

The exclusion criterion is:

1. Child not at home after 3 attempts

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22815 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Malaria prevalence | Measured one time in randomly selected participants at baseline and 6, 12, 18 and 24 months post intervention deployment.
  The primary outcome of the study will be malaria parasite prevalence (any plasmodium species) in participants aged 1-15 years old

SECONDARY OUTCOMES:
Prevalence of parasitaemia in children aged 1-5 years | Measured one time in randomly selected participants at baseline and 6, 12, 18 and 24 months post intervention deployment.
  Proportion of children aged 1-5 years with blood smears positive for parasites by microscopy at the time of community cross-sectional surveys.
Prevalence of parasitaemia in children aged 6-10 years | Measured one time in randomly selected participants at baseline and 6, 12, 18 and 24 months post intervention deployment.
  Proportion of children aged 6-10 years with blood smears positive for parasites by microscopy at the time of community cross-sectional surveys.
Prevalence of parasitaemia in children aged 11-15 years | Measured one time in randomly selected participants at baseline and 6, 12, 18 and 24 months post intervention deployment.
  Proportion of children aged 11-15 years with blood smears positive for parasites by microscopy at the time of community cross-sectional surveys.
Prevalence of anaemia in children under 5 years | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of children under 5 years of age with haemoglobin < 11 g/dL at the time of community cross-sectional surveys.
Proportion of households that owned at least one LLIN | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of households with at least one long-lasting insecticidal net (LLIN) at the time of community cross-sectional surveys.
Proportion of households with at least one LLIN for every two occupants | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of households with at least one long-lasting insecticidal net (LLIN) per every two household occupants at the time of community cross-sectional surveys.
Proportion of household residents who slept under an LLIN the previous night | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of household residents who report sleeping under a long-lasting insecticidal net (LLIN) the previous night at the time of community cross-sectional surveys.
LASER intervention coverage | Measured at 6, 12, 18 and 24 months post initial intervention deployment
  Proportion of sampled households in the LASER intervention arm that have the required number of SCJ Guardian spatial emanators present at the time of community cross-sectional surveys.
Indoor residual spraying (IRS) coverage | Measured at 6, 12, 18 and 24 months post inital intervention deployment
  Proportion of surveyed households that report received indoor residual spraying (IRS) as part of the study in the IRS arm.
Malaria incidence in patients of all ages from health facility surveillance | Data captured monthly for 24 months post intervention deployment
  Number of cases of malaria diagnosed at participating health facilities among patients of all ages residing in study clusters per unit time, divided by the estimated population of the cluster villages.
Anopheles spp. vector density | Measured at baseline and 6, 12, 18 and 24 months post initial intervention deployment
  Number of female Anopheles mosquitoes collected by ultra violet light traps per household at the time of entomology surveys in randomly selected households
Anopheles mosquitoes species composition | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of each Anopheles mosquito species identified among collected specimens at the time of entomology surveys by molecular identification.
Sporozoite rate in Anopheles spp. mosquitoes | Measured at baseline and 6, 12, 18 and 24 months post initial intervention deployment
  Proportion of screened Anopheles mosquitoes that test positive for Plasmodium sporozoites.
Insecticide resistance in Anopheles spp. | Measured at baseline and 6, 12, 18 and 24 months post initial intervention deployment
  Proportion of Anopheles mosquitoes surviving standard WHO insecticide susceptibility tests at the time of entomology surveys.
Frequency of insecticide resistance genetic variants in Anopheles mosquitos | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of screened Anopheles mosquitoes carrying molecular markers associated with insecticide resistance at the time of entomology surveys.
Acceptability of LASER and preventive measures by participant demographics | Baseline, 12 months post intervention deployment and within 3 months post intervention withdrawal
  Proportion of participants reporting acceptability of spatial repellents (SR) and other preventive measures, assessed using structured questionnaires. Data stratified by gender, age group, and socio-economic activity categories.
Appropriateness of LASER and other preventive measures in local context | Baseline, 12 months post intervention deployment, and within 3 months post intervention withdrawal.
  Proportion of participants rating long-acting spatial emanators (LASER) and other preventive measures as appropriate for their local context, assessed using structured questionnaires. Stratified by gender, age group, and socio-economic activity.
Proportion of participants reporting barriers to LASER use | Baseline, 12 months post intervention deployment, and within 3 months post intervention withdrawal.
  Proportion of participants in LASER arm identifying specific barriers to LASER intervention use, assessed using semi-structured interviews and focus group discussions. Barriers categorized and quantified by thematic analysis.
Reasons for non-adherence to LASER intervention | Baseline, 12 months post intervention deployment, and within 3 months post intervention withdrawal.
  Proportion of non-adherent participants citing specific reasons for non-adherence, assessed using semi-structured interviews. Reasons categorized by thematic analysis and reported as percentage of non-adherent participants per category.
Contextual factors affecting LASER delivery and transferability | Baseline, 12 months post intervention deployment, and within 3 months post intervention withdrawal.
  Number and type of contextual factors (social, environmental, health system) affecting LASER delivery identified through key informant interviews and focus group discussions. Factors categorized by thematic analysis to inform transferability to other malaria endemic areas.
Cost per household protected per year | Cost data collected monthly throughout 24-month trial period; final calculation at 24 months post intervention deployment
  Annual cost in US dollars (USD) per household protected by the interventions, calculated as total intervention costs divided by the number of households receiving protection. Costs include implementation, distribution, and maintenance costs.
Incremental cost-effectiveness ratio: Cost per malaria case averted | 24 months post intervention deployment
  Incremental cost in US dollars (USD) per malaria case averted compared to standard of care.
Incremental cost-effectiveness ratio: Cost per DALY averted | 24 months post intervention deployment
  Incremental cost in US dollars (USD) per disability-adjusted life year (DALY) averted compared to standard of care
Mean Household Willingness to Pay | 24 months post intervention deployment
  Mean willingness to pay in US dollars (USD) and local currency units (LCU) per household for the intervention, assessed using contingent valuation methodology with bidding game administered via structured questionnaire.
Budget impact at scale | 24 months post intervention deployment
  Estimated total cost in US dollars (USD) for scaling up the intervention to a defined target population, calculated using budget impact analysis modeling based on observed unit costs and projected coverage scenarios.
Equity of intervention coverage | Measured at baseline and 6, 12, 18 and 24 months post intervention deployment
  Proportion of sampled households that have the intervention present at the time of community cross-sectional surveys assessed as coverage by socio-economic status group (quantile).

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI Center for Global Health Research, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes